CLINICAL TRIAL: NCT04036539
Title: Evaluation of the Effects of Photobiomodulation on Orthodontic Movement of Molar Verticalization With Mini-implant: a Randomized Double-blind Protocol Study
Brief Title: Photobiomodulation on Molar Verticalization With Mini-implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, PhD, clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: verticalization
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2020-01

CONDITIONS: Orthodontic Appliances; Low-Level Light Therapy
Keywords: orthodontic treatment,; photobiomodulation,; mini-implant,; verticalization of molars

STUDY DESIGN:
Intervention Model Description: 34 individuals will be randomly divided into 2 groups: G1 (control group) - verticalization by mini-implant + PBM simulation (placebo); G2 (experimental group) - verticalization by mini-implant + PBM.
Who Masked: Participant, Investigator
Masking Description: Only one external research collaborator, with dental training, who will be responsible for the treatments (which will open the envelopes of randomization), will know which photobiomodulation treatment will be assigned to each patient. The identification of each group will be revealed by this collaborator to all involved only after statistical analysis of the data. Therefore, the researcher responsible for data collection, and the statistician will be blinded to the treatments assigned to the groups. The patient will also be blind to the type of treatment performed since the mini-implant placement treatment will be identical in both groups and the laser treatment for photobiomodulation will be simulated in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (placebo) (Placebo Comparator): Patients in Control will receive the photobiomodulation placebo,application, but with the laser off. Procedures will be performed immediately after the application of forces (placement of elastic bandages) on the tooth, as described: Simulations will be performed with the same laser.This will require 10 seconds of application simulation per point. As 10 points will be simulated, it will take 100 seconds for this simulation.5 points lingual and 5 points at vestibular
  Interventions: Procedure: Placement of the mini-implant and verticalization
- Experimental: (Experimental): Experimental: Molar verticalization + PBM (n = 17 + 3) - patients will receive laser treatment (photobiomodulation) in order to modulate orthodontic movement and act on inflammation and pain. The procedures will be performed immediately after the application of forces (placement of elastic bandages) on the tooth, as described:The irradiations will be performed with the red diode laser ( = 660 nm) with 100 milliwatts output power The power of the device will be 100miliWatts and the wavelength used will be 808 nanometers (± 10nm). The optical fiber diameter of the device is 600 micrometer, therefore a spot (area) of 0.002826 centimeter2. The energy delivered per point will be 1Joule. This will require 10 seconds of application per point. As 10 points will be irradiated, the total application time will be 100 seconds and the total energy delivered will be 10Joule. The energy density will be 25 Joule / cm2 and the power density will be 35.38 Watt / cm2
  Interventions: Procedure: Placement of the mini-implant and verticalization

INTERVENTIONS:
Procedure: Placement of the mini-implant and verticalization — an orthodontic mini-implant will be installed in the retromandibular region. The site will be anesthetized. The region will be pre-drilled by about 5mm with a spear drill attached to an implant motor. Once the mini-implant has been selected, it will be locked into position using a kit-specific digital key. Being threaded clockwise until the intramucosal mini-implant is at the gingival level. After installation, a metallic orthodontic lingual will be glued to the molar mesial to be verticalized. The lingual button will be glued to the inclined molar mesial with orthodontic adhesive. A gray chain elastomeric ligature will attach the head of the mini-implant to the lingual button glued to the molar mesial. A light force of 150gr will be imposed (measured with a tensiometer) in all cases, regardless of tooth position. This chain elastic will be changed every 30 days for a period of 3 months. After 90 days of the experiment time, the mini-implants will be removed.

SUMMARY:
The objective of this study will be to evaluate the effect of photobiomodulation on the acceleration of the orthodontic movement of molar verticalization and its effect on pain and inflammation of the periodontal tissues.

Thirty-four healthy patients aged 30-60 years, who need to recover the prosthetic space for oral rehabilitation after loss of the posterior inferior dental elements and inclination of the adjacent element, will be randomly divided into 2 groups: G1 (control group) - verticalization by mini-implant + PBM (photobiomodulation) simulation (placebo); G2 (experimental group) - verticalization by mini-implant + PBM. The movements will occur with the aid of mini-implants and elastomeric chains ligatures. The PBM will occur with diode laser application, 660 nm (nanometers), 100mW (milliwatts), receiving 1J(joule) per point, 10s (seconds), 10 points (5 per buccal and 5 per lingual) and radiant exposure of 25 J / cm². The crevicular gingival fluid (FGC) will be collected to analyzed Interleukins IL1β, IL-6, IL-8, IL-10(Interleukins) and TNF-α (tumor necrosis factor) by ELISA (enzyme-linked immunosorbent assay). Radiographic shots will be taken each month to ascertain the amount (in degrees) of verticalization. To evaluate the pain, the Visual Analogue Scale will be used in all the consultations, and to evaluate the quality of life, the OHIP-14 (oral health impact profile) questionnaire will be applied. Analgesics will be given and the number of drugs will be counted. If the data are normal, they will be submitted to the Student's t-test. The data will be presented as means ± SD(standard deviation) and the value of p will be defined as <0.05.

DETAILED DESCRIPTION:
Loss of a dental element can generate several repercussions in the stomatognathic system. According to the latest survey by the Ministry of Health, in 2010, Brazilian adults had, on average, 7 missing teeth. This loss may lead to movement of the adjacent teeth and the antagonist, which would make prosthetic rehabilitation harder to do. Anchoring systems, such as mini-implants, have been increasingly used as a treatment option because they act with heavy but controlled forces and without side effects. Recent studies have shown that photobiomodulation (PBM) can accelerate orthodontic movement in the molar intrusion. The objective of this study will be to evaluate the effect of photobiomodulation on the acceleration of the orthodontic movement of molar verticalization and its effect on pain and inflammation of the periodontal tissues.

Thirty-four healthy patients aged 30-60 years, who need to recover the prosthetic space for oral rehabilitation after loss of the posterior inferior dental elements and inclination of the adjacent element, will be randomly divided into 2 groups: G1 (control group) - verticalization by mini-implant + PBM simulation (placebo); G2 (experimental group) - verticalization by mini-implant + PBM. The movements will occur with the aid of mini-implants and elastomeric chains ligatures. The PBM will occur with diode laser application, 660 nm, 100mW, receiving 1J per point, 10s, 10 points (5 per buccal and 5 per lingual) and radiant exposure of 25 J / cm². The orthodontic forces of verticalization (corresponding to any exchange of elastomeric ligation) will be applied every 30 days and the PBM will be applied immediately, 3 and 7 days of each month, for a period of 3 months. The crevicular gingival fluid (FGC) will be collected on the 1st, 3rd and 7th days after the first activation, and then on the 3rd day of the following two months. Interleukins IL1β, IL-6, IL-8, IL-10 and TNF-α will be analyzed by ELISA. Radiographic shots will be taken each month to ascertain the amount (in degrees) of verticalization. To evaluate the pain, the Visual Analogue Scale will be used in all the consultations, and to evaluate the quality of life, the OHIP-14 questionnaire will be applied. Analgesics will be given and the number of drugs will be counted. If the data are normal, they will be submitted to the Student's t-test. The data will be presented as means ± SD and the value of p will be defined as <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree and sign the informed consent
* healthy (ASA I - negative medical history),
* systolic blood pressure less than 140mmHg and diastolic blood pressure less than 90mmHg,
* heart rate with 70 ± 20 beats / minute
* requiring oral rehabilitation after loss of some posterior lower dental element (1st molar),
* with favorable periodontal condition to the installation of mini-implants. Any questions during the research period should be informed to the researcher so that the researcher can take the appropriate measures (the latter should provide some form of personal contact).

Exclusion Criteria:

* Patients who are latex allergic,
* pregnant or breastfeeding,
* smokers,
* diabetics,
* patients undergoing head and neck radiotherapy,
* coagulation disorders requiring antibiotic prophylaxis for placement of mini-implants, with absolute indication for use of local anesthetics with vasoconstrictors,
* with decompensated systemic disease,
* with systemic or local infection (periodontitis or periodontal abscess),
* who have used anti-inflammatory drugs in the last 3 months before orthodontic treatment.
* Patients who may have any complications during the research period, such as allergic reactions to any of the materials used, allergic reaction to paracetamol®,

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Radiographic measurements | through study completion on average of one year
  Radiographic measurements to assess movement rate through tooth angulation versus time at baseline, 30, 60 and 90 days after treatment, Movement rate - With the aid of a ruler (Morelli, Sorocaba, SP, Brazil) and a protractor (transparent Waleu 10290001®), radiographic measurements will be taken at baseline, 30, 60 and 90 days to ascertain the amount (in degrees) of verticalization, using as reference the line of the occlusal plane and the long axis of the inclined tooth (García, 2017). These measurements will be recorded in degrees in each patient's chart for further analysis.

SECONDARY OUTCOMES:
Pain during movement: Visual Analog Scale (VAS) | through study completion on average of one year
  Assess pain during orthodontic verticalization movement using the Visual Analog Scale (VAS) at baseline 30, 60, and 90 days after mini-implant placement Pain during movement - Will be assessed by applying the visual analog scale (VAS) with a 100 mm line, with both ends closed. One end has the indication "0" and the other "100" which means "no pain" and "unbearable pain" respectively. Marking instructions will always be given to the patient by the same operator. Each patient will be instructed to mark with a vertical stroke the point that best corresponds to the pain intensity at the moment of evaluation
Assess the amount of painkillers ingested | through study completion on average of one year
  Assess the amount of painkillers ingested in the period to verify that this therapy is effective in reducing pain during baseline orthodontic movement, 3 and 7 days, 30, 60, and 90 days after mini-implant placement.
  Rescue medication - Another parameter analyzed will be the amount of analgesics ingested. At the beginning of the research, a paracetamol® (drug with purely analgesic effect card will be delivered to each patient. It should be stored until the end and its use will be released only in case of pain. At the end of the experiment, the number of pills will be evaluated as another parameter to measure pain.
Oral health-related quality of life (HRQoL): OHIP-14 | through study completion on average of one year
  Oral health-related quality of life (HRQoL) will be assessed using the OHIP-14 baseline questionnaire and 90 days after treatment Analysis of oral health-related quality of life (Oral health impact profile questionnaire - Ohip-14) - This questionnaire is a simplified form of the original OHIP-49 questionnaire. Ohip-14 will be used to assess the impact of oral health on the quality of life of research participants. Ohip-14 is used to measure perceived needs. It measures the impact of oral changes on oral health related quality of life. The participant will answer 14 questions by giving their answers the values 0 (never), 1 (almost never), 2 (sometimes), 3 (most of the time) and 4 (always).

CONTACTS AND LOCATIONS:
Overall Officials: Anna carolina RT Horliana, Phd, Principal Investigator — University of Nove de Julho
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernandes MRU, Suzuki SS, Suzuki H, Martinez EF, Garcez AS. Photobiomodulation increases intrusion tooth movement and modulates IL-6, IL-8 and IL-1beta expression during orthodontically bone remodeling. J Biophotonics. 2019 Oct;12(10):e201800311. doi: 10.1002/jbio.201800311. Epub 2019 Jul 8. PMID 31001928
- [Result] Schalch TO, Palmieri M, Longo PL, Braz-Silva PH, Tortamano IP, Michel-Crosato E, Mayer MPA, Jorge WA, Bussadori SK, Pavani C, Negreiros RM, Horliana ACRT. Evaluation of photodynamic therapy in pericoronitis: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2019 Apr;98(17):e15312. doi: 10.1097/MD.0000000000015312. PMID 31027098
- [Result] Bauer HC, Duarte FL, Horliana AC, Tortamano IP, Perez FE, Simone JL, Jorge WA. Assessment of preemptive analgesia with ibuprofen coadministered or not with dexamethasone in third molar surgery: a randomized double-blind controlled clinical trial. Oral Maxillofac Surg. 2013 Sep;17(3):165-71. doi: 10.1007/s10006-012-0360-7. Epub 2012 Sep 5. PMID 22949122